CLINICAL TRIAL: NCT01066806
Title: Efficacy of Optimal Levels of Dietary Dairy on Modulation of Adolescent Weight
Brief Title: Adequate Dairy Intake on Weight Change in Girls
Acronym: DQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Joan Lappe, Professor of Medicine, Creighton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-14739
Record Dates: First submitted 2010-01-19; First posted 2010-02-10 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high calcium diet (Experimental)
  Interventions: Behavioral: counseling on increasing calcium intake
- normal calcium diet (Active Comparator)
  Interventions: Other: observation

INTERVENTIONS:
Behavioral: counseling on increasing calcium intake — The American Academy of Pediatrics recommends that adolescents ingest at least four servings of dairy food and at least 1300 mg calcium per day.
  Arms: high calcium diet
Other: observation — observe normal dairy intake
  Arms: normal calcium diet

SUMMARY:
SPECIFIC AIM The aim of this study is to determine if increasing calcium intake to recommended levels with dairy foods in adolescent females with habitually low calcium intake and above-the-median body mass index (BMI) for sex and age will decrease body fat gain compared to similar females who continue their low calcium intake. .

HYPOTHESIS Post-menarcheal adolescent girls with habitually low calcium intake who consume dairy foods providing at least 1200 mg of calcium per day will have a smaller increase in percent body fat, as measured by dual energy absorptiometry, during one year than post-menarcheal adolescent girls on a usual diet of 600 mg of calcium per day or less.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-14 years old (must be this age when consent is signed)
* Above the 50th percentile for BMI
* Above the 85th percentile for BMI with approval from their primary physician
* At least one and one- half years post menarche
* Habitual dietary calcium intake of 600mg/d or less as assessed by 3 day diet diary. This will be inclusive of supplemental calcium and dietary intake.
* Willingness to increase dietary calcium (low fat [skim, 1%, 2%] milk or yogurt) for one year

Exclusion Criteria:

* Menarche prior to age 10
* History of lactose intolerance or milk allergy
* Weight >300 pounds
* BMI > 97 percentile for age and gender
* Pregnancy
* Chronic disease or disorder like diabetes, polycystic ovarian syndrome, thyroid disease, seizures or cancer (cancer is ok if it has been >10 years)
* Use of steroids like prednisone, prednisolone, hydrocortisone, Flovent, Advair, or Nasonex
* Use of weight reducing medications like Meredia, alli, Dexatrim or Xenical
* Use of contraceptives like Yasmin, Ortho Tri-Cyclen, Apri, Aviane or Depo-Provera for any reason, including acne (see inclusive list)
* Use of acne medications like Accutane or high dose Vitamin A
* Use of ADHD medications like Adderall, Ritalin, Concerta. (Per Dr. Ramaswamy-Straterra OK) (see inclusive list)
* Use of seizure medications like Lamictal or Phenobarb (see inclusive list)
* Use of anti-depressants like Prozac or Effexor (see inclusive list)
* Diagnosed eating disorder
* Dieting behavior with weight loss > 10 pounds in the last 3 months (IF YES, consult with Project Manager)
* Metal in the skeleton (pins, rods, etc)
* Sibling of a child who is or has been on a dietary study in the last 5 years
* Total body BMC Z-score below -2.0 at baseline
* Participating in other ongoing research protocols

Ages: 13 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2008-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
percent change in body fat | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Lappe, PhD, Principal Investigator — Creighton University, Osteoporosis Research Center
Locations (1):
- Creighton University Medical Center, Osteoporosis Research Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Lappe JM, McMahon DJ, Laughlin A, Hanson C, Desmangles JC, Begley M, Schwartz M. The effect of increasing dairy calcium intake of adolescent girls on changes in body fat and weight. Am J Clin Nutr. 2017 May;105(5):1046-1053. doi: 10.3945/ajcn.116.138941. Epub 2017 Mar 15. PMID 28298396